CLINICAL TRIAL: NCT06355817
Title: Distraction Techniques in Periocular Anesthesia: Tapping vs Vibration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Winnipeg Regional Health Authority (Other)
Responsible Party: Principal Investigator, Yen Minh Cung, MD, Principle Investigator, University of Manitoba
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HS25941
Record Dates: First submitted 2024-03-28; First posted 2024-04-09 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Anesthetics, Local; Blepharoplasty; Age-Related Ptosis; Adult; Humans; Lidocaine; Ophthalmologic Surgical Procedure; Vibration; Surgery
Keywords: Study, Crossover; Pain Measurement; Prospective Study

STUDY DESIGN:
Intervention Model Description: Each patient will receive both interventions and serve as their own comparator.
Who Masked: Participant, Care Provider
Masking Description: The participant and surgeon was not made aware of which intervention the participant would receive first until the time of the procedure. Randomization was made at the time of the procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Tap then Vibrate (Active Comparator): Tapping for the first eye/side during infiltration of local anesthetic, then vibration for the second eye.
  Interventions: Device: Vibration; Other: Tapping
- Group B: Vibrate then Tap (Experimental): Vibration first, then tapping
  Interventions: Device: Vibration; Other: Tapping

INTERVENTIONS:
Device: Vibration — Vibration Assist Device, held to the forehead
  Other Names: Facial Massager
Other: Tapping — Tapping on the forehead

SUMMARY:
To compare the efficacy of topical tapping vs vibration in lowering pain scores for periocular anesthesia injections.

DETAILED DESCRIPTION:
Participants will be selected from 3 local oculoplastics surgeons' procedural slates during the study period. Eligible participants are those who will be undergoing bilateral eye procedures. They will be randomized into one of two groups: Group A will receive tapping on their forehead for their first eye injection of local anesthesia, and then vibration to their forehead for the second eye. Group B will receive the reverse. Pain scores will be aggregated and an average taken to help determine which method is superior. The vibration assist device (variety of facial massagers are available on Amazon for roughly $16-20CDN) is being considered in addition to the current standard of tapping or no tactile distraction at all during the injection of local anesthetic. The 11-point pain Visual Analog Scale will be used to help grade pain experience after each eye is frozen. To help qualify, if there is a difference, the patient will be asked if they felt one technique was better than the other by a little, quite a bit, or a lot.

ELIGIBILITY:
Inclusion Criteria:

* adult patients undergoing elective bilateral eye procedures such as blepharoplasty

Exclusion Criteria:

* previous eyelid surgery
* inability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-09-21 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-03-19 (Actual)

PRIMARY OUTCOMES:
Pain Reduction in Tapping vs Vibration distraction techniques in peri-ocular local anesthesia | Immediately after both eyes receive local anesthetic
  How effective each intervention was in reducing the pain of peri-ocular local anesthesia, as graded on an 11-point Visual Analog Pain Scale (from 0-10 where 10/10 pain is the worst and 0/10 pain is no pain at all)

SECONDARY OUTCOMES:
Difference in Pain Reduction | Immediately after both eye receive local anesthetic
  If there was a difference, subjective qualitative grading of how much difference: a little bit, quite a bit, or a lot

CONTACTS AND LOCATIONS:
Overall Officials: Yen Minh Cung, MD, Principal Investigator — University of Manitoba, Dept of Ophthalmology
Locations (1):
- Misericordia Health Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
After 5 years the hard copies of data collection sheets and master list will be shredded.

REFERENCES:
- [Background] Gostimir M, Hussain A. A Systematic Review and Meta-analysis of Methods for Reducing Local Anesthetic Injection Pain Among Patients Undergoing Periocular Surgery. Ophthalmic Plast Reconstr Surg. 2019 Mar/Apr;35(2):113-125. doi: 10.1097/IOP.0000000000001209. PMID 30664129
- [Background] Aminabadi NA, Farahani RM, Balayi Gajan E. The efficacy of distraction and counterstimulation in the reduction of pain reaction to intraoral injection by pediatric patients. J Contemp Dent Pract. 2008 Sep 1;9(6):33-40. PMID 18784857
- [Background] Strazar AR, Leynes PG, Lalonde DH. Minimizing the pain of local anesthesia injection. Plast Reconstr Surg. 2013 Sep;132(3):675-684. doi: 10.1097/PRS.0b013e31829ad1e2. PMID 23985640
- [Background] Babamiri K, Nassab R. The evidence for reducing the pain of administration of local anesthesia and cosmetic injectables. J Cosmet Dermatol. 2010 Sep;9(3):242-5. doi: 10.1111/j.1473-2165.2010.00503.x. PMID 20883298
- [Background] Govas P, Kazi R, Slaugenhaupt RM, Carroll BT. Effect of a Vibratory Anesthetic Device on Pain Anticipation and Subsequent Pain Perception Among Patients Undergoing Cutaneous Cancer Removal Surgery: A Randomized Clinical Trial. JAMA Facial Plast Surg. 2019 Dec 1;21(6):480-486. doi: 10.1001/jamafacial.2019.0733. PMID 31513234
- [Background] Ing EB, Philteos J, Sholohov G, Kim DT, Nijhawan N, Mark PW, Gilbert J. Local anesthesia and anxiolytic techniques for oculoplastic surgery. Clin Ophthalmol. 2019 Jan 10;13:153-160. doi: 10.2147/OPTH.S188790. eCollection 2019. PMID 30666086
- [Background] Melzack R, Wall PD. Pain mechanisms: a new theory. Science. 1965 Nov 19;150(3699):971-9. doi: 10.1126/science.150.3699.971. No abstract available. PMID 5320816
- [Background] Chen BK, Eichenfield LF. Pediatric anesthesia in dermatologic surgery: when hand-holding is not enough. Dermatol Surg. 2001 Dec;27(12):1010-8. doi: 10.1046/j.1524-4725.2001.01854.x. PMID 11849262
- [Background] Smith KC, Comite SL, Balasubramanian S, Carver A, Liu JF. Vibration anesthesia: a noninvasive method of reducing discomfort prior to dermatologic procedures. Dermatol Online J. 2004 Oct 15;10(2):1. PMID 15530291
- [Background] McKinlay JR, Hofmeister E, Ross EV, MacAllister W. EMLA cream-induced eye injury. Arch Dermatol. 1999 Jul;135(7):855-6. doi: 10.1001/archderm.135.7.855. No abstract available. PMID 10411170
- [Background] Reed ML. Surgical pearl: mechanoanesthesia to reduce the pain of local injections. J Am Acad Dermatol. 2001 Apr;44(4):671-2. doi: 10.1067/mjd.2001.110641. No abstract available. PMID 11260545
- [Background] Katz J, Melzack R. Measurement of pain. Surg Clin North Am. 1999 Apr;79(2):231-52. doi: 10.1016/s0039-6109(05)70381-9. PMID 10352653
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Result] Fayers T, Morris DS, Dolman PJ. Vibration-assisted anesthesia in eyelid surgery. Ophthalmology. 2010 Jul;117(7):1453-7. doi: 10.1016/j.ophtha.2009.11.025. Epub 2010 Mar 19. PMID 20303597
- [Result] Sharma P, Czyz CN, Wulc AE. Investigating the efficacy of vibration anesthesia to reduce pain from cosmetic botulinum toxin injections. Aesthet Surg J. 2011 Nov;31(8):966-71. doi: 10.1177/1090820X11422809. Epub 2011 Oct 14. PMID 22001341
- See also: Specific vibration assist device used in the study — https://www.amazon.com/Bar-Massager-T-Shape-Electric-Sensitive/dp/B074PQM987/ref=sr_1_2?crid=14B17OMO2MX8B&keywords=beauty+bar&qid=1673905519&sprefix=beauty+bar%2Caps%2C181&sr=8-2